CLINICAL TRIAL: NCT04840238
Title: A Multicentre, Phase-II, Randomised, Double Blind, Placebo-controlled Study to Assess the Safety and the Efficacy of a Weekly Administered Dose of 30,000 IU Vitamin D (Colecalciferol) in Deficient Patients Diagnosed With PCOS
Brief Title: 30000 IU Per Week Vitamin D Treatment in PCOS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: Pharma Patent Kft. (Unknown)
Responsible Party: Principal Investigator, Istvan Takacs, M.D., DSc., Director of Department, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAT15-PCODD
Record Dates: First submitted 2020-07-14; First posted 2021-04-09 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Polycystic Ovary Syndrome; Vitamin D Deficiency
MeSH Terms: conditions — Polycystic Ovary Syndrome; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cholecalciferol (Experimental): Cholecalciferol 30,000IU weekly orally
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): Placebo tablets weekly orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — 30,000IU cholecalciferol
  Arms: Cholecalciferol
Drug: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
This is a human, II/b phase, multicentre, randomised, double blind, placebo-controlled study to assess the safety and the efficacy of a weekly administered dose of 30,000 IU vitamin D (colecalciferol) in deficient patients diagnosed with PCOS.

Investigational products: 30.000 IU vitamin D or placebo administered once a week for 12-weeks-long period, followed by a 12-week-long open label treatment 30.000 IU vitamin D in a follow-up period.

Each participant should be checked for regular dietary Ca intake and to assure the optimal calcium level the supplementation is provided with a commercially available Citrocalcium 200 mg tablets.

Setting:

I. Baseline and screening period:

Baseline period considered as when the exogenous Vitamin D intake should not exceed the level of 1000 IU intake per day or a total 5000 NE per week dosages applied (in forms of any Vitamin D3 medication or multivitamin products) at least for 30 days prior the assessment made.

II. Double-blind treatment period:

Once a week per os applied Vitamin D or placebo treatment for 12 weeks according to randomisation of trial subjects in a 1:1 assignment. By the end of this period an interim assessment will be performed based on the analysis of primary efficacy parameters, stratification to responder and non-responder groups.

III. Open label and follow-up phase:

An open-label 30000 IU of Vitamin D treatment on weekly basis. (Vitamin D3 Pharma Patent 30000 IU tablets) for additional 12 weeks and continue with the follow-up assessments. A compassionate use of patient diary for additional 26 weeks.

Objectives:

Primary objectives: to assess the efficacy as a recovery of ovarian function based on progesterone levels and menses diary in at least 20% of trial subjects, compared to placebo treated group Secondary Objectives: assess the efficacy and safety of orally administered vitamin D treatment by the changes in 25(OH) D levels in PCOS patients.

Explore the changes in Ovarian-morphology based on the results of standard TVUS Imaging: detection of adverse drug reactions during treatment periods, by frequency and distribution compared to follow-up periods and placebo group.

Anticipated participants: 168

ELIGIBILITY:
Inclusion Criteria:

* Female subject age >18 years.
* Clinical and/or biochemical hyperandrogenism and the proven PCOS by the "Rotterdam" criteria, (ovarian dysfunction, oligo- and/or anovulation, and the morphology of polycystic ovaries on ultrasound images when other etiologies are excluded)
* 25(OH)D levels are between 10-28 ng/ml by inclusion
* Subject can not be under any kind of ongoing hormone or metformin therapies and no indication that requires continuation
* Has the ability and willingness to understand and comply with study procedures and to give written informed consent prior to enrollment in the study or initiation of study procedures
* Study subject has the ability and willingness to understand and comply with study procedures and to give written informed consent prior to enrollment in the study or initiation of study procedures

Exclusion Criteria:

* Has been exposed to any investigational agent within 3 month of enrolment to the study
* Sever metabolic disease on endocrine disease in etiology different from PCOS
* Significant obesity (BMI> 36)
* Any other signs of lab results that may lead to other etiologies in differentiation, or menopause
* Increased serum calcium level results or symptoms of hypercalcemia in last one year
* Hypercalciuria or kidney stone appearance in last one year
* Sever kidney diseases (CKD 3 or higher)
* Chronic or serious disease, which can significantly influence the absorption, metabolism of vitamin D or Ca
* Heart failure or angina pectoris,
* More than 1000 IU vitamin D per day intake or in total >5000 IU per week within 1 month prior to trial (in any forms medication, or nutritional food supplement). The patient is not under hormonal therapy for ovulation stimulation purposes and was not involved in two months prior the study
* The patient is under hormonal therapy for the aim of ovulation stimulation or was involved in within 3 months prior the study
* Existence or suspected gravidity
* Any other finding or symptoms which are by the opinion of the Investigator may indicate a potential interference with the safety of participating trial subjects
* Has a known hypersensitivity to any of the investigational drug or vehicle components.
* Concomitant medication which is not allowed:

  * glycosides
  * metformin
  * magnesium-containing preparations (antacids)
  * cholestyramine and other ion exchange resins, orlistat
  * thiazide diuretics
  * regular use of microsomal enzyme inducers (anticonvulsants, sedatives, etc.).
  * corticosteroids (except for dermatological use)
  * products containing phosphorus
  * regular use of laxatives (such as paraffin oil)
  * fat absorption inhibitory drugs
  * any kind of hormone therapy (including therapeutic use of birth control pills, within 2 months prior inclusion) except treatment of stabile hypothyroidism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Polycystic ovarian syndrome develops in only females
Enrollment: 115 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Recovery of ovarian function | Up to 32 weeks, continuously
  Recovery of ovarian function is detected by changes in progesterone levels (lutal phase progesterone level reaches 2 ng/ml)

SECONDARY OUTCOMES:
Length of menstrual cycle | Up to 32 weeks
  Determined by patient reported number of days between two menstrual cycles
Variation in menstrual cycles length | Up to 32 weeks
  Determined by patient reported menstrual cycle length and regularity, measured in days
Incidence of adverse events | Up to 32 weeks, continuously
  Incidence of adverse events (safety and tolerability), evaluated at every visit
Change in serum calcium level | Up to 32 weeks, continuously
  Change in serum calcium levels in mmol/l (safety measure), evaluated every clinical visit
Change in urinary calcium/creatinine ratio | Up to 32 weeks
  Change in urinary calcium/creatinine ratio ([mmol/l]/[umol/l]) (safety measure), evaluated every clinical visit
25(OH)D levels | Up to 32 weeks
  Evaluation of treatment of changes in 25(OH)D blood levels compared between treatment groups
Change in fasting glucose level | Up to 32 weeks
  Change in fasting glucose level (mmol/l), measured at every visit
Change in hemoglobin A1c level | Up to 32 weeks
  Change in hemoglobin A1c level (IFCC validated, mmol/mol), measured every 12 weeks
Change in ovarian morphology | Up to 32 weeks
  Changes in ovarian follicle count assessed by TVUS and evaluated by the Rotterdam criteria (having 12 or more follicles, measuring between 2 and 9 mm)

CONTACTS AND LOCATIONS:
Overall Officials: István Takács, MD, DSc., Principal Investigator — Semmelweis University - Dept. of Medicine and Oncology
Locations (8):
- Hungary (8):
  - Semmelweis University - Departement Medicine and Oncology, Budapest
  - MediMOM Healthy Center, Budapest
  - Róbert Károly Hospital, Budapest
  - Gynpraxis Nőgyógyászat, Debrecen
  - Somogy County Kaposi Mór Teaching Hospital, Kaposvár
  - Borsod-Abaúj-Zemplén County Hospital, Miskolc
  - SZTE-ÁOK - 1st Dept. of Internal MEdicine, Szeged
  - Gynofarm Outpatient Clinic, Székesfehérvár

IPD SHARING:
Plan to Share IPD: No